CLINICAL TRIAL: NCT03655860
Title: Evaluation of SIMEOX on Flow and Volume Elicited in Healthy Subjects
Brief Title: Effects of SIMEOX on Flow and Volume
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never started, was replaced by NCT04150601
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIMEOX-01; 2018/08AOU/312 (Other: CEHF)
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIMEOX (Experimental): Use of the device SIMEOX to exhale
  Interventions: Device: SIMEOX

INTERVENTIONS:
Device: SIMEOX — SIMEOX is a device generating a succession of gentle depression at the mouth.

SUMMARY:
This study will investigate the effects of the SIMEOX (an airway clearance device) on flow and volume generated in healthy subjects

DETAILED DESCRIPTION:
This is a pilot study assessing the effect of the SIMEOX device on flow and volume generated in healthy subjects.

Assessment of flow and volume will be performed before and during the application of the SIMEOX. Vital capacity and expiratory flow will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the instructions

Exclusion Criteria:

* Obesity (BMI > 30kg/m²)
* Active smoker
* Severe scoliosis
* Cardiovascular ou neuromuscular disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Change in expiratory volume | 5min
  Expiratory volume before and during the use of the SIMEOX will be compared
Change in expiratory volume flow rate | 5min
  Expiratory flow rate before and during the use of the SIMEOX will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Grégory Reychler, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- William Poncin, Brussels, Belgium